CLINICAL TRIAL: NCT03713840
Title: Community Partnering to Encourage Healthy Beverage Intake Through Child Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Anisha Patel, Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-07599
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Obesity
Keywords: nutrition; child care; obesity
MeSH Terms: conditions — Obesity | interventions — Child Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Beverages in Child Care (Experimental): Child care centers in the experimental arm received 12-week intervention that promoted consumption of healthy beverages (water, unsweetened low-fat milk) and discouraged consumption of unhealthy beverages (juice, sugar-sweetened beverages, high-fat or sweetened milk). The multi-pronged intervention was delivered via child care centers, targeted children, parents, and child care staff, and included education, environmental changes, and policies.
  Interventions: Behavioral: Healthy Beverages in Child Care
- Control (No Intervention): Child care centers in the control arm received access to intervention materials at a later date.

INTERVENTIONS:
Behavioral: Healthy Beverages in Child Care — 12-week intervention promoted consumption of healthy beverages (water, unsweetened low-fat milk) and discouraged consumption of unhealthy beverages (juice, sugar-sweetened beverages, high-fat or sweetened milk). The multi-pronged intervention was delivered via child care centers, targeted children, parents, and child care staff, and included education, environmental changes, and policies.
  Arms: Healthy Beverages in Child Care

SUMMARY:
Beverage consumption is an important determinant of young children's weight, yet few obesity prevention interventions focus comprehensively on encouraging healthy beverage consumption. This quasi-experimental study evaluated whether a childcare-based intervention, combining environmental changes, education/promotion, and policy supports to promote healthy beverage intake, improved at-home beverage consumption and weight status among children ages 2-5 years.

DETAILED DESCRIPTION:
Inappropriate intake of whole milk, fruit juice, and sugar-sweetened beverages is associated with childhood obesity, obesity-related co morbidities, and dental caries, yet there are few proven interventions to promote child intake of healthy beverages consistent with national guidelines. Child care facilities provide a potential venue for influencing healthy beverage intake in children and families. The overall objective of this study is to use principles of community-based participatory research (CBPR; an approach in which researchers partner with community members to conduct research) to develop, pilot test, and examine the acceptability, feasibility, sustainability, and preliminary outcomes of a child care-based intervention to encourage child intake of age-appropriate, guideline-recommended beverages. The central hypothesis is that a multi-level intervention consisting of educational strategies to encourage intake of guideline-recommended beverages; increased accessibility of lead-free, fluoridated, drinking water in child care and at home; and evidence-based child care and home beverage policies will lead to healthier beverage intake and reduced childhood obesity. This hypothesis was tested through a quasi-experimental trial in four child care centers. Centers were randomized to a control (delayed-intervention) condition or to receive a 12-week intervention that promoted consumption of healthy beverages (water, unsweetened low-fat milk) and discouraged consumption of unhealthy beverages (juice, sugar-sweetened beverages, high-fat or sweetened milk). The multi-pronged intervention was delivered via child care centers, targeted children, parents, and child care staff, and included education, environmental changes, and policies. Outcomes were measured at baseline and immediately post-intervention and included children's (n =154) at-home beverage consumption (assessed via parental report) and overweight/obese weight status (assessed via objectively measured height and weight).

ELIGIBILITY:
Inclusion Criteria:

1. Child care centers were eligible if they were in San Mateo County, CA, were licensed, had enrolled at least ten children ages 2-5 years, participated in the Child and Adult Care Food Program (CACFP: a federal nutrition assistance program providing funding for meals and snacks), had English or Spanish-speaking staff, and served primarily English or Spanish-speaking families.
2. Two to five-year-old children were eligible if they were enrolled in participating child care facilities.
3. Parents of eligible children were able to participate in beverage intake surveys if they spoke English or Spanish.

Exclusion Criteria:

1. Non-center, unlicensed, and higher-income child care facilities were ineligible to participate.
2. Parents unable to speak Spanish/English were excluded.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2013-08-15 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-01 (Actual)

PRIMARY OUTCOMES:
BMI (kg/m2) | 12 weeks
  Height and weight measurements were obtained per NHANES anthropometry procedures manual. Weight in kilograms was divided by height in meters squared to obtain BMI.
BMI% | 12 weeks
  We computed age and sex specific BMI% using the Centers for Disease Control and Prevention age- and sex-specific growth curves
Proportion obese | 12 weeks
  BMI% greater than or equal to 95% comprised obesity; The proportion of children meeting that definition was obtained
Proportion overweight | 12 weeks
  BMI% greater than or equal to 85% comprised obesity; The proportion of children meeting that definition was obtained

SECONDARY OUTCOMES:
SSB intake (ounces/day) | 12 weeks
  Intake of sugar-sweetened beverages (SSBs) or beverages with added sugar was obtained using 24 hour recalls
Water intake (ounces/day) | 12 weeks
  Intake of water was obtained using 24 hour recalls
Low fat/skim milk intake (ounces/day) | 12 weeks
  Intake of low fat (1%) or skim milk was obtained using 24 hour recalls
2%/whole milk intake (ounces/day) | 12 weeks
  Intake of 2% or whole milk was obtained using 24 hour recalls
100% fruit juice (ounces/day) | 12 weeks
  Intake of 100% fruit juice was obtained using 24 hour recalls

CONTACTS AND LOCATIONS:
Overall Officials: Anisha Patel, MD, MSPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No